CLINICAL TRIAL: NCT02665884
Title: Diurnal Fluctuations of Intraocular Pressure in EX-Press Valve Blebs in Glaucoma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0085-15-HYMC
Record Dates: First submitted 2015-11-29; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-11

CONDITIONS: GLAUCOMA
MeSH Terms: conditions — Glaucoma | interventions — Intraocular Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Glaucoma EX-PRESS: Glaucoma patients who underwent glaucoma surgery between the years 2014-2015 and had diurnal intraocular pressure measurements over 24 hours.
  Interventions: Other: Intraocular Pressure Measurement
- Control Group: Glaucoma patients who had been treated with anti-glaucoma drops and had diurnal intraocular pressure measurements over 24 hours.
  Interventions: Other: Intraocular Pressure Measurement

INTERVENTIONS:
Other: Intraocular Pressure Measurement — Diurnal fluctuations of intraocular pressure will be measured and compared

SUMMARY:
Diurnal fluctuations of intraocular pressure in EX-Press Valve Blebs in Glaucoma Patients

Intraocular pressure (IOP) reduction is the mainstay of glaucoma management. (1) Open-angle glaucoma (OAG) is generally managed by decreasing the intraocular pressure (IOP) to a level that the physician believes will prevent further glaucomatous damage. However, in a significant proportion of patients, the visual fields continue to deteriorate in spite of office pressures within the range of normal values (8). It has been suggested that the progressive damage in some cases could be caused by peaks of IOP or diurnal IOP variability not detected by tonometry during office hours. It is possible that certain drugs or surgical interventions are more effective than others in dampening these fluctuations. The purpose of our study is to compare the diurnal IOP fluctuations in glaucoma patients treated with medications or Ex-press filtration surgery.

DETAILED DESCRIPTION:
Diurnal fluctuations of intraocular pressure in EX-Press Valve Blebs in Glaucoma Patients

Department of Ophthalmology, Hillel-Yaffe Medical Center, affiliated with the Bruce Rappaport School of Medicine, The Technion, Haifa, Israel

Introduction:

Intraocular pressure (IOP) reduction is the mainstay of glaucoma management. (1) Medication alone is sometimes not sufficient to reduce excessively high IOP, and pharmaceutical intolerance may develop or damage can occur to the optic nerve, warranting surgical intervention. (2) The filtering bleb is considered to be the cornerstone of IOP control after glaucoma filtration surgery drainage device implantation. (3) It enables the flow of the aqueous humor from the anterior chamber to the subconjunctiva, episclera, sclera and choroid, thereby lowering the IOP. (4-6) Filtration and drainage devices, such as the EX-Press device (Alcon Laboratories, Fort Worth, Texas, USA), offer a surgical alternative to glaucoma medical therapy. (7) Open-angle glaucoma (OAG) is generally managed by decreasing the intraocular pressure (IOP) to a level that the physician believes will prevent further glaucomatous damage. However, in a significant proportion of patients, the visual fields continue to deteriorate in spite of office pressures within the range of normal values (8). It has been suggested that the progressive damage in some cases could be caused by peaks of IOP or diurnal IOP variability not detected by tonometry during office hours. (9, 10) In another study, Asrani et al. (11) showed that IOP fluctuations are an independent risk factor in patients with glaucoma and as such may need to be treated specifically. It is possible that certain drugs or surgical interventions are more effective than others in dampening these fluctuations. The purpose of our study is to compare the diurnal IOP fluctuations in glaucoma patients treated with medications or Ex-press filtration surgery.

Materials and Methods The study will include 20 open-angle glaucoma (OAG) patients underwent Ex-Press filtration surgery, and 20 OAG patients treated with medications alone. All patients will have 12 IOP measurements with 2 hours interval, starting at 10 AM until 10 AM of the following morning.

ICARE® PRO tonometer (Icare Finland Oy, Espoo, Finland) will be used for the measurement of IOP. The rebound motion of its light weighted probe will be recorded during contact of the probe with the cornea. (12, 13) The rate of deceleration of the probe is a function of IOP. The ICARE® PRO has a built-in inclination sensor that allows downward measurement of the eye in the supine position as well as in the normal upright sitting position. ICARE® PRO allows for measurement of IOP in the seated and supine positions. During IOP recording, patients will be supine or upright, and the tip of the probe will be applied perpendicular to the cornea. Two markers engraved on the piston of the probe indicated its ideal positioning. The reliability of the measurement is displayed on the ICARE® PRO tonometer screen and guided our measurements.

Fluctuations in IOP will be compared between the Ex-press filtration surgery eye and the fellow (intra-group comparison). Inter-group comparison of IOP fluctuation will be performed between the Ex-press filtration surgery eye and medically treated eye of different patients.

ELIGIBILITY:
Inclusion Criteria: .

* Glaucoma patients that underwent EX-PRESS surgery

Exclusion Criteria:

* Angle closure glaucoma
* Neovascular glaucoma
* High refractive error

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 20 open-angle glaucoma (OAG) patients underwent Ex-Press filtration surgery, and 20 OAG patients treated with medications alone.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of diurnal fluctuations of intraocular pressure | One year
  Comparison of diurnal fluctuations of intraocular pressure in glaucoma patients with and without EX-Press valve surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] The Advanced Glaucoma Intervention Study (AGIS): 7. The relationship between control of intraocular pressure and visual field deterioration.The AGIS Investigators. Am J Ophthalmol. 2000 Oct;130(4):429-40. doi: 10.1016/s0002-9394(00)00538-9. PMID 11024415
- [Result] Watson PG. When to operate on open angle glaucoma. Eye (Lond). 1987;1 ( Pt 1):51-4. doi: 10.1038/eye.1987.8. PMID 2881812
- [Result] Levene RZ. Glaucoma filtering surgery: factors that determine pressure control. Ophthalmic Surg. 1984 Jun;15(6):475-83. PMID 6462607
- [Result] Picht G, Grehn F. Classification of filtering blebs in trabeculectomy: biomicroscopy and functionality. Curr Opin Ophthalmol. 1998 Apr;9(2):2-8. doi: 10.1097/00055735-199804000-00002. PMID 10180508
- [Result] Hu CY, Matsuo H, Tomita G, Suzuki Y, Araie M, Shirato S, Tanaka S. Clinical characteristics and leakage of functioning blebs after trabeculectomy with mitomycin-C in primary glaucoma patients. Ophthalmology. 2003 Feb;110(2):345-52. doi: 10.1016/S0161-6420(02)01739-6. PMID 12578779
- [Result] DeBry PW, Perkins TW, Heatley G, Kaufman P, Brumback LC. Incidence of late-onset bleb-related complications following trabeculectomy with mitomycin. Arch Ophthalmol. 2002 Mar;120(3):297-300. doi: 10.1001/archopht.120.3.297. PMID 11879132
- [Result] Netland PA, Sarkisian SR Jr, Moster MR, Ahmed II, Condon G, Salim S, Sherwood MB, Siegfried CJ. Randomized, prospective, comparative trial of EX-PRESS glaucoma filtration device versus trabeculectomy (XVT study). Am J Ophthalmol. 2014 Feb;157(2):433-440.e3. doi: 10.1016/j.ajo.2013.09.014. Epub 2013 Nov 7. PMID 24210765
- [Result] Kidd MN, O'Connor M. Progression of field loss after trabeculectomy: a five-year follow-up. Br J Ophthalmol. 1985 Nov;69(11):827-31. doi: 10.1136/bjo.69.11.827. PMID 4063249
- [Result] DRANCE SM. DIURNAL VARIATION OF INTRAOCULAR PRESSURE IN TREATED GLAUCOMA. SIGNIFICANCE IN PATIENTS WITH CHRONIC SIMPLE GLAUCOMA. Arch Ophthalmol. 1963 Sep;70:302-11. doi: 10.1001/archopht.1963.00960050304004. No abstract available. PMID 14048787
- [Result] Zeimer RC, Wilensky JT, Gieser DK, Viana MA. Association between intraocular pressure peaks and progression of visual field loss. Ophthalmology. 1991 Jan;98(1):64-9. doi: 10.1016/s0161-6420(91)32340-6. PMID 2023735
- [Result] Asrani S, Zeimer R, Wilensky J, Gieser D, Vitale S, Lindenmuth K. Large diurnal fluctuations in intraocular pressure are an independent risk factor in patients with glaucoma. J Glaucoma. 2000 Apr;9(2):134-42. doi: 10.1097/00061198-200004000-00002. PMID 10782622
- [Result] Iliev ME, Goldblum D, Katsoulis K, Amstutz C, Frueh B. Comparison of rebound tonometry with Goldmann applanation tonometry and correlation with central corneal thickness. Br J Ophthalmol. 2006 Jul;90(7):833-5. doi: 10.1136/bjo.2005.089870. Epub 2006 May 3. PMID 16672330
- [Result] Martinez-de-la-Casa JM, Garcia-Feijoo J, Castillo A, Garcia-Sanchez J. Reproducibility and clinical evaluation of rebound tonometry. Invest Ophthalmol Vis Sci. 2005 Dec;46(12):4578-80. doi: 10.1167/iovs.05-0586. PMID 16303951